CLINICAL TRIAL: NCT03079141
Title: Study on Half-dose Photodynamic Therapy Versus Eplerenone in Chronic CenTRAl Serous Chorioretinopathy (SPECTRA Trial)
Brief Title: Photodynamic Therapy Versus Eplerenone: Treatment Trial for Chronic Central Serous Chorioretinopathy
Acronym: SPECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, CJFBoon, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P16.255
Record Dates: First submitted 2017-03-02; First posted 2017-03-14 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Chronic Central Serous Chorioretinopathy
MeSH Terms: interventions — Eplerenone; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Half-dose photodynamic therapy (PDT) (Active Comparator): In the PDT treatment arm, all patients will receive an intravenous drip through which half-dose (3 mg/m2) verteporfin (Visudyne®) is administered, with an infusion time of 10 minutes. At exactly 15 minutes after the start of the infusion, PDT laser treatment is performed with standard 50 J/cm2 fluency, a wavelength of 689 nm, and a treatment duration of 83 seconds.
  When patients are randomized to the PDT arm of this study, they will receive this treatment as a first cCSC treatment. Moreover, PDT can be performed in patients in whom SRF is still present on OCT at the Evaluation Visit at 3 months after the start of eplerenone treatment.
  Interventions: Other: Photodynamic therapy
- Oral eplerenone treatment (Active Comparator): Patients will receive 25 milligrams oral eplerenone once daily for a week, and - when no abnormalities during blood testing for potassium and renal clearance can be detected both before treatment and during the first week of treatment - will receive 50 milligrams oral eplerenone for another 11 weeks thereafter.
  When patients are randomized to the eplerenone arm of this study, they will receive this treatment as a first cCSC treatment. Moreover, eplerenone treatment can be initiated in patients in whom SRF is still present on OCT at the Evaluation Visit at 3 months after PDT treatment.
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Patients will receive 25 milligrams oral eplerenone once daily for a week, and - when no abnormalities during blood testing for potassium and renal clearance can be detected both before treatment and during the first week of treatment - will receive 50 milligrams oral eplerenone for another 11 weeks thereafter.
  When patients are randomized to the eplerenone arm of this study, they will receive this treatment as a first cCSC treatment. Moreover, eplerenone treatment can be initiated in patients in whom SRF is still present on OCT at the Evaluation Visit at 3 months after PDT treatment.
  Other Names: Inspra
  Arms: Oral eplerenone treatment
Other: Photodynamic therapy — In the PDT treatment arm, all patients will receive an intravenous drip through which half-dose (3 mg/m2) verteporfin (Visudyne®) is administered, with an infusion time of 10 minutes. At exactly 15 minutes after the start of the infusion, PDT laser treatment is performed with standard 50 J/cm2 fluency, a wavelength of 689 nm, and a treatment duration of 83 seconds.
  When patients are randomized to the PDT arm of this study, they will receive this treatment as a first cCSC treatment. Moreover, PDT can be performed in patients in whom SRF is still present on OCT at the Evaluation Visit at 3 months after the start of eplerenone treatment.
  Arms: Half-dose photodynamic therapy (PDT)

SUMMARY:
Chronic central serous chorioretinopathy (cCSC) is a relatively frequently occurring eye disease that is often diagnosed in patients in the professionally active age range. In this disease, a subretinal fluid accumulation occurs, due to abnormalities in both the choroid and the retinal pigment epithelium. This specific form of macular degeneration can cause permanent vision loss, image distortion, and loss of color and contrast vision. An early diagnosis and treatment may improve the visual outcome and quality of life.

To date there is no international consensus on the optimal treatment of cCSC. Many retrospective studies suggest that treatment with photodynamic therapy (PDT) is effective in chronic CSC. Treatment with oral eplerenone may also be effective in this disease.

In this proposed prospective randomized controlled trial, cCSC patients will be randomized into one of both treatment groups: either half-dose PDT or oral eplerenone treatment. The trial is a superiority study, because retrospective studies suggest that PDT treatment may be more effective than eplerenone treatment.

The null hypothesis of the study is that PDT treatment is more effective than eplerenone treatment in patients with active cCSC. The alternative hypothesis is that PDT treatment is not superior to eplerenone treatment.

Treatment success will not only be based on characteristics on ophthalmological imaging, but also on functional endpoints (both on the outcome of questionnaires, best-corrected visual acuity, and microperimetry), which are most important from a patient's perspective.

The study will take place in 3 large tertiary referral university hospitals in The Netherlands that have extensive experience with conducting clinical trials (Academic Medical Center (Amsterdam, the Netherlands), Radboud University Medical Center (Nijmegen, the Netherlands), and Leiden University Medical Center (Leiden, the Netherlands). Both the Radboud University Medical Center and the Leiden University Medical Center have been involved in the first prospective randomized controlled trial that is currently conducted in cCSC.

This study will last 2 years per participant. Each participant will visit the outpatient clinic for a maximum number of 6 visits.

A total number of 107 patients will be included in the trial. Depending on the speed of inclusion of patients in this trial, the total duration of this study can be determined.

DETAILED DESCRIPTION:
Chronic central serous chorioretinopathy (cCSC) is a relatively frequently occurring eye disease that is often diagnosed in patients in the professionally active age range. In this disease, a subretinal fluid accumulation occurs, due to abnormalities in both the choroid and the retinal pigment epithelium. This specific form of macular degeneration can cause permanent vision loss, image distortion, and loss of color and contrast vision. An early diagnosis and treatment may improve the visual outcome and quality of life.

To date there is no international consensus on the optimal treatment of cCSC. Many retrospective studies suggest that treatment with photodynamic therapy (PDT) is effective in chronic CSC. Treatment with oral eplerenone may also be effective in this disease.

In this proposed prospective randomized controlled trial, cCSC patients will be randomized into one of both treatment groups: either half-dose PDT or oral eplerenone treatment. The trial is a superiority study, because retrospective studies suggest that PDT treatment may be more effective than eplerenone treatment.

The null hypothesis of the study is that PDT treatment is more effective than eplerenone treatment in patients with active cCSC. The alternative hypothesis is that PDT treatment is not superior to eplerenone treatment.

Treatment success will not only be based on characteristics on ophthalmological imaging, but also on functional endpoints (both on the outcome of questionnaires, best-corrected visual acuity, and microperimetry), which are most important from a patient's perspective.

The study will take place in 3 large tertiary referral university hospitals in The Netherlands that have extensive experience with conducting clinical trials (Academic Medical Center (Amsterdam, the Netherlands), Radboud University Medical Center (Nijmegen, the Netherlands), and Leiden University Medical Center (Leiden, the Netherlands). Both the Radboud University Medical Center and the Leiden University Medical Center have been involved in the first prospective randomized controlled trial that is currently conducted in cCSC.

This study will last 2 years per participant. Each participant will visit the outpatient clinic for a maximum number of 6 visits, depending on the outcome of treatment. Study evaluations will be mostly part of regular clinical care.

A total number of 107 patients will be included in the trial. Depending on the speed of inclusion of patients in this trial, the total duration of this study can be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥ 18 years of age and able to give written informed consent;
* Active chronic central serous chorioretinopathy (cCSC);
* Subjective visual loss > 6 weeks, interpreted as onset of active disease;
* Foveal subretinal fluid (SRF), on optical coherence tomography (OCT), at Baseline Examination;
* ≥1 ill-defined hyperfluorescent leakage areas on fluorescein angiography (FA) with retinal pigment epithelial window defect(s) that are compatible with cCSC;
* Hyperfluorescent areas on indocyanine green angiography (ICGA).

Exclusion Criteria:

* Any previous treatments for active CSC;
* Previous prescription of mineralocorticoid receptor antagonists, for cCSC or for other diseases;
* Current treatment with corticosteroids (topical or systemic), corticosteroid use within 3 months before possible start of trial treatment, or anticipated start of corticosteroid treatment within the first 2 years from the start of the trial period;
* Evidence of another diagnosis that can explain serous SRF or visual loss;
* Best-corrected visual acuity < 20/200 (Snellen equivalent);
* Profound chorioretinal atrophy in central macular area on ophthalmoscopy and OCT;
* Myopia > 6D;
* Visual loss and/or serous detachment on OCT < 6 weeks;
* Continuous and/or progressive visual loss > 18 months or serous detachment on OCT > 18 months;
* No hyperfluorescence on ICGA;
* Intraretinal edema on OCT;
* (relative) Contraindications for FA or ICGA;
* (relative) Contraindications for photodynamic treatment (pregnancy, porphyria, severely disturbed liver function). Pregnancy will not be routinely tested in female patients, but the possibility of pregnancy will be discussed during screening
* (relative) Known contraindications for initiation of eplerenone treatment (hyperkalemia, abnormal renal clearance, severe hepatic insufficiency (Child-Pugh C), type 2 diabetes mellitus with microalbuminuria, concomitant use of potassium supplements, potassium-sparing diuretics, strong CYP3A4 inhibitors, or the combination of an ACE-inhibitor and an angiotensin receptor blocking agent). Pregnancy will not be routinely tested in female patients, but the possibility of pregnancy will be discussed during screening;
* Soft drusen in treated eye or fellow eye, signs of choroidal neovascularization on ophthalmoscopy and/or FA/ICGA of the study eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Absence of subretinal fluid on OCT scan | 3 months after (start) of treatment
  Absence of subretinal fluid on OCT scan

SECONDARY OUTCOMES:
Macular sensitivity on microperimetry | At evaluation visits during study, depending on the effect of treatment. All patients will visit the outpatient clinic at 3 months, at 1 year, and at 2 years after the (start of) treatment.
  Macular sensitivity on microperimetry
Mean change in best-corrected visual acuity | At evaluation visits during study, depending on the effect of treatment. All patients will visit the outpatient clinic at 3 months, at 1 year, and at 2 years after the (start of) treatment.
  Mean change in Early Treatment of Diabetic Retinopathy Study best-corrected visual acuity
Vision-related quality of life as reported on the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) | At evaluation visits during study, depending on the effect of treatment. All patients will visit the outpatient clinic at 3 months, at 1 year, and at 2 years after the (start of) treatment.
  Vision-related quality of life as reported on the National Eye Institute Visual Function Questionnaire (NEI-VFQ-25)
Number of cross-over treatments needed in each treatment arm | During study. At the evaluation visit at 3 months after the (start of) treatment, a possible cross-over treatment can be performed.
  Number of cross-over treatments needed (half-dose photodynamic therapy to eplerenone treatment, and vice versa) in each treatment arm
The long-term outcome both after successful treatment and after non-successful treatment | One year and two year after (start of) therapy
  Persistent absence of subretinal fluid on OCT
The number of (S)AEs in the 2 different treatment groups. | At the several evaluation visits within the study, at 3 months, at 1 year, and at 2 years after (the start of) treatment
  The number of (S)AEs in the 2 different treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Camiel JF Boon, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (3):
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen

IPD SHARING:
Plan to Share IPD: No
No plan.

REFERENCES:
- [Derived] Feenstra HMA, Diederen RMH, Lamme MJCM, Tsonaka R, Fauser S, Yzer S, van Rijssen T, Gkika T, Downes SM, Schlingemann RO, Hoyng CB, van Dijk EHC, Boon CJF. INCREASING EVIDENCE FOR THE SAFETY OF FOVEA-INVOLVING HALF-DOSE PHOTODYNAMIC THERAPY FOR CHRONIC CENTRAL SEROUS CHORIORETINOPATHY. Retina. 2023 Mar 1;43(3):379-388. doi: 10.1097/IAE.0000000000003686. Epub 2023 Jan 2. PMID 36727801